CLINICAL TRIAL: NCT00185991
Title: Comparison of Once Daily Versus 8 Hour Dosing of Gentamicin for the Treatment of Intrapartum Chorioamnionitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Yasser Yehia El-Sayed, Stanford University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 80104
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Chorioamnionitis
MeSH Terms: conditions — Chorioamnionitis | interventions — Gentamicins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Once daily Gentamicin (Active Comparator)
  Interventions: Drug: gentamicin
- Every eight hour Gentamicin (Active Comparator)
  Interventions: Drug: gentamicin

INTERVENTIONS:
Drug: gentamicin — Daily gentamicin (5 mg/kg intravenously, then placebo doses IV after 8 and 16 hours).
  Eight hour gentamicin (2 mg/kg intravenously, then 1.5 mg/kg IV after 8 and 16 hours).

SUMMARY:
To compare once daily versus 8 hour dosing of gentamicin for the treatment of chorioamnionitis.

ELIGIBILITY:
Inclusion Criteria:

- clinical diagnosis of chorioamnionitis

Exclusion Criteria:

- maternal renal disease, intrauterine fetal death, allergy to gentamicin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2004-06; Primary Completion 2006-10 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Afebrile at 24 hours and no endometritis | 24 hours after delivery

SECONDARY OUTCOMES:
Neonatal outcomes | Time of delivery to time of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Yehia El-Sayed, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Lyell DJ, Pullen K, Fuh K, Zamah AM, Caughey AB, Benitz W, El-Sayed YY. Daily compared with 8-hour gentamicin for the treatment of intrapartum chorioamnionitis: a randomized controlled trial. Obstet Gynecol. 2010 Feb;115(2 Pt 1):344-349. doi: 10.1097/AOG.0b013e3181cb5c0e. PMID 20093909